CLINICAL TRIAL: NCT06502730
Title: Nursing Led Interventions: Effect of Creating Opportunities for Parent Empowerment Program on Mother- Infant Interaction, Sense of Competence and Mental Health Outcome.
Brief Title: COPE Program , Mental Health, Mother- Infant Interaction, Sense of Competence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matrouh University (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Principal Investigator, Seham El-Sayed Saleh Hassan, Assistant Professor of pediatric nursing, faculty of nursing, Matrouh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AU-20-4-248
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Empowerment; Competence; Outcome; Interaction
Keywords: COPE;; Maternal Competence;; Maternal Mental Health;; Parent-Infant Interaction;; Preterm neonates
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Mothers of preterm neonates who will not receive COPE program.
- Study group (Experimental): Mothers of preterm neonates who will receive COPE program.
  Interventions: Behavioral: Creating Opportunities for Parent Empowerment (COPE) Program

INTERVENTIONS:
Behavioral: Creating Opportunities for Parent Empowerment (COPE) Program — It helps to recognize the critical role of parents and encourage taking an active role in their neonate's care, engaging in dyadic interaction with their neonate. COPE program consists of two types of educational information; as teaching parents about normal physical, developmental and behavioral characteristics of their preterm infants and the best ways to interact with them and facilitate their development.
  Arms: Study group

SUMMARY:
The aim of the study is to:

- Evaluate the effect of creating opportunities for parent empowerment program on maternal sense of competence, mental health outcome and mother-infant interaction.

RESEARCH HYPOTHESES

* Mothers of preterm neonates who receive creating opportunities for parent empowerment program exhibit high level of competence than those who don't.
* Mothers of preterm neonates who receive creating opportunities for parent empowerment program exhibit less stress level than those who don't.
* Mothers of preterm neonates who receive creating opportunities for parent empowerment program exhibit high interaction than those who don't.

The mothers of preterm neonates will be assigned into two equal groups as follows:

* Study group (group II) mothers of preterm neonates who will receive COPE program.
* Control group (group I) mothers of preterm neonates who will not receive COPE program.

DETAILED DESCRIPTION:
* Research Design: A quasi-experimental (pre-posttest) research design will be used.
* Setting: The study will be conducted at the Neonatal Intensive Care Unit at Smouha Specialty Hospital in Alexandria.
* Subjects: A convenience sampling of 60 mothers of preterm infants who admitted to the previously mentioned setting
* During the 1st day of preterm admission to NICU data concerning characteristics of neonates and their mothers' in both groups will be obtained from medical records using tool I.
* The pretest will be conducted to the mothers of neonates on the 1st day of admission in the NICU to assess mothers' sense of competence and perceived stress by interviewing them to collect data using tool II, III and mother infant interaction in both groups by observation using tool IV.
* After completion of the pretest, the mothers in the study group will receive COPE program, then at the 7th day of the study posttest will be done for both group

ELIGIBILITY:
Inclusion Criteria:

* The mother age more than 20 years, educated and has no experience of premature birth
* The mother has no postpartum discomforts (such as, bleeding, depression or pain
* Premature neonates( gestational age 37 weeks)
* Birth weight < 2500 g or > 1500 g (LBW)
* Five-minute Apgar score > 7
* Neonate not with any medically restricted conditions (e.g., intraventricular hemorrhage or intracerebral hemorrhage (grades III and IV).
* Neonate not on ant ventilation assisted devices, such as ventilator or CPAP

Exclusion Criteria:

-

Ages: 34 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Parenting Sense of Competency Scale (PSOC) | 7 days
  This scale was developed by Gibaud-Wallston & Wandersman, 1978, the Chinese version of the PSOC Scale (C-PSOC) to assess the mothers' sense of competence and satisfaction with parenting. The C-PSOC includes 17 items.
Modified Parental Stressor Scale (PSS): NICU | 7 days
  This scale was developed by (Miles et al. 1993). It is used to assess perceived stress of mothers with preterm infants during the NICU hospitalization of their infant. The PSS:NICU is a 50-item self-report scale that measures parental stress related to four dimensions of the NICU environment: sights and sounds in the NICU (5 items); the infant's appearance (21 items); staff behaviors and communication (13 items), and parent interaction with baby (11 items).
Parent-Infant Interaction Observation (PIIO) Checklist: | 7 days
  It is an observational Scale developed by (Svanberg, et al., 2013), It is a screening tool for parent-infant interactions for infant aged from 0-6 months. It includes 13 interactional items such as: Infant positioning, eye contact, vocalizations, affect engagement and synchrony, warmth and affection, holding and handling, verbal commenting (mind- mindedness), attunement/ harmony to distress, bodily intrusiveness, expressed expectations, empathic understanding, responsive turn taking, and baby's self-soothing strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Seham Saleh, Principal Investigator — Matrouh University
Locations (1):
- Matrouh university, Marsá Maţrūḩ, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibaud-Wallston J, Wandersman LP. Parenting sense of competence scale. 1978. https://researchingparents.wordpress.com/2013/02/15/parentingsense- of-competence-psoc/
- [Background] Jnaneswari. K, Dr. Manjubala Dash. Effect of COPE Program (Creating Opportunities for Parent Empowerment) on Maternal Stress and Parent Neonate Interaction among NICU Mothers. Archives of Reproductive Medicine and Sexual Health. 2020; 3(1): 16-23.
- [Background] Miles MS, Funk SG, Carlson J. Parental Stressor Scale: neonatal intensive care unit. Nurs Res. 1993 May-Jun;42(3):148-52. PMID 8506163
- [Background] P.O. Svanberg, J. Barlow & W. Tigbe (2013) The Parent-Infant Interaction Observation Scale: reliability and validity of a screening tool, Journal of Reproductive and Infant Psychology, 31:1, 5-14, DOI: 10.1080/02646838.2012.751586